CLINICAL TRIAL: NCT01706640
Title: An Open- Label,Multicentre, Observational, Prospective, Real-time Data Capturing of Usage, Outcome & Physician Satisfaction of Coseal in Cardio- Vascular- Thoracic Operative and Re- Operative Procedures
Brief Title: An Open Label,Observational, Real Time Data Capturing of Usage & Outcome of Coseal
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medanta, The Medicity, India (Other)
Responsible Party: Principal Investigator, Dr. Ali Zamir Khan, Head of Department, Minimally Invasive & Robotic Thoracic Surgery, Medanta, The Medicity, India
Other Study IDs: MM/CTVS/2012/001
Record Dates: First submitted 2012-10-08; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is Open- Label, Observational, Prospective, Real-time data capturing of Usage, Outcome & Physician satisfaction of Coseal in Cardio- Vascular-Thoracic Operative and Re- Operative procedures.

Objective of this study is to assess current practice pattern and best practice sharing of usage of Coseal by collecting data on (1) Sealing suture lines along arterial and venous reconstruction(2) Patients undergoing cardiac surgery to prevent or reduce the incidence, severity and extent of post surgical adhesion enforcement of suture lines in lung resection procedures (3) From this data to document and generate a real life experience on the use of Coseal in cardio vascular and thoracic surgery.

Number of expected patient enrollment is 750 from 20 participating sites.

DETAILED DESCRIPTION:
Objectives:

* Assessing current practice pattern and best practice sharing of usage of Coseal as per IFU by collecting data on oSealing suture lines along arterial and venous reconstructions oPatients undergoing cardiac surgery to prevent or reduce the incidence, severity and extent of post surgical adhesion enforcement of suture and staple lines in lung resection procedures
* From this data to document and generate a real life experience on the use of Coseal in cardio vascular and thoracic surgery
* To possibly create a guideline for usage of Sealant in routine practice in India
* To study delivery methods and clinical impact in minimally invasive surgery like VATS and robotic surgery

End points

Primary Endpoint

1. Cardio vascular sealing:

   To report the effectiveness and safety of COSEAL in the control of anastomotic suture line and needle hole suture bleeding during vascular reconstruction by checking the incidence of immediate anastomotic sealing and the presence of persistent intra-operative and postoperative bleeding average time to achieve hemostasis for a single bleeding site after 60 s of clamping without manual compression In case of sternotomy, Hemostasis time in mns, which is operative time comprised between the removal of cardio-pulmonary bypass cannulae and the closure of the sternum.

   Overall postoperative bleeding in mL/m² revision for bleeding Minor complications, major complications, mortality
2. Efficacy of Coseal in prevention or reduction of adhesion in re-do surgeries for patients with staged operations for congenital cardiac malformation re-operated on during the follow-up period of the registry

   Incidence of adhesions. location and extension of adhesion by measuring the percentage of surface affected for each of the following regions: pericardial or retrosternal, inferior or diaphragmatic region, right lateral or atrial region, region around the great vessels, pulmonary surface.

   Overall evaluation (dissection easy or difficult) Incidence of subjects free of adhesions.

   Severity (at each of these sites, the adhesions will be graded as follows:

   absence of adhesion; 1: filmy and avascular; 2: dense and/or vascular; and 3: cohesive)
3. Air leak: incidence of immediate (at the time of closure) and prolonged post-operative air leak, Use in redo surgery for air leak.

Secondary Endpoints

1. Cardiovascular (sealing and adhesion prevention):

   1. Total operative time
   2. Nature and duration of first operation
   3. Nature and duration of redo operation, and time for dissection from sternotomy to end of dissection for prevention of adhesions )
   4. Length of intensive care stay
   5. Length of hospital stay
   6. Infection rate
   7. Quality of wound healing
   8. Quality of life (SF36)
2. Thoracic and Lung

   1. Sealing the suture/ staple line on table Use of buttressing
   2. Total operative time
   3. Drain output
   4. Drain duration
   5. Length of hospital stay
   6. Prolonged air leak (more than 5 days) (>5 days is the new standard for prolonged aire leak accepted in 2011 by the EU Soc of CVTS, see ref.)
   7. Infection rate
3. In all cases,

   1. intra and post-operative blood loss
   2. FFP, Transfusion
   3. Reoperation for bleeding purpose
4. Others

   1. Surgeons satisfaction
   2. Easiness of product handling during application (VAS)

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiovascular and thoracic surgery who require use of Coseal as a treatment strategy.
2. Patient undergoing open, Video Assisted surgery and robotic surgery to be included and analysed as subgroups
3. Written informed consent obtained from the patient or legal representative for data collection post surgery in patients who had Coseal used intraoperatively (data privacy laws).

Exclusion Criteria:

1. Known hypersensitivity to components of the investigational product
2. Known Immune system disorders, immunodeficiency
3. Concomitant use of any other anti-adhesion product
4. Concurrently participating in another clinical trial and having received another investigational drug or device within the last 30 days
5. Unplanned re-operation in case of use for anti-adhesion
6. Contraindications for use of Coseal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient falling under inclusion criteria can take part in to bthe study
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-11 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Cardio Vascular Outcome | 18 months
  To report the effectiveness and safety of COSEAL in the control of anastomotic suture line and needle hole suture bleeding during vascular reconstruction by checking the incidence of immediate anastomotic sealing and the presence of persistent intra-operative and postoperative bleeding

SECONDARY OUTCOMES:
Cardiovascular (sealing and adhesion prevention): | 18 months
  To Capture total operative time,nature and duration of first operation,nature and duration of redo operation, and time for dissection from sternotomy to end of dissection for prevention of adhesions )
Thoracic and Lung (Sealing and Adhesion prevention) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ali Z Khan, MS,FRCS,FRCS, Principal Investigator — Medanta, The Medicity
Locations (1):
- Medanta, The Medicity, Gurgaon, Haryana, India